CLINICAL TRIAL: NCT04619316
Title: Enhancing Radioiodine Incorporation Into Radio Iodine Refractory Thyroid Cancers With MAPK Inhibition: A Single Center Pilot Study
Brief Title: Enhancing Radioiodine Incorporation Into Radio Iodine Refractory Thyroid Cancers With MAPK Inhibition
Acronym: ERRITI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, PD Dr. med. Wolfgang Fendler, Principal Investigator, University Hospital, Essen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERRITI; 2016-002941-49 (EudraCT Number); Version 2.0 (Other: Sponsor)
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — trametinib; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRAF wild type (Other): In BRAF wild type patients trametinib 2mg (1-0-0) is applied daily over a time span of 3 weeks, then the effect is evaluated via 123I whole-body scintigraphy
  Interventions: Drug: Trametinib 2 MG [Mekinist]
- BRAF V600E Mutation (Other): In BRAF wild type patients trametinib 2mg (1-0-0) and dabrafenib 75mg (2-0-2) are applied daily over a time span of 3 weeks, then the effect is evaluated via 123I whole-body scintigraphy
  Interventions: Drug: Trametinib 2 MG [Mekinist] and Dabrafenib 75 MG (2-0-2) [Tafinlar]

INTERVENTIONS:
Drug: Trametinib 2 MG [Mekinist] — Monotherapy with Trametinib is given in patients with BRAF wildtype.
  Arms: BRAF wild type
Drug: Trametinib 2 MG [Mekinist] and Dabrafenib 75 MG (2-0-2) [Tafinlar] — Combination therapy is given in patients with BRAF V600E mutation.
  Arms: BRAF V600E Mutation

SUMMARY:
This is a prospective interventional trial that aims to restore iodine incorporation in tumoral lesions of patients with unresectable, radioiodine-refractory thyroid cancer.

DETAILED DESCRIPTION:
This is a prospective interventional study testing the hypothesis that the inhibition of MEK can restore iodine incorporation in BRAF wild type (WT) and a combined inhibition of BRAF and MEK can restore iodine incorporation in BRAFV600E mutant (MUT), radioiodine-refractory (RAIR) thyroid cancer. Patients with proven iodine negative tumor lesion(s) will be included in this study. Patients will then receive Trametinib (WT-group) or Dabrafenib and Trametinib combination-therapy (MUT-group) for approximately 3 weeks, after which a Thyrogen-stimulated 123I SPECT imaging will be performed. For patients whose tumor(s) demonstrate sufficient iodine incorporation in the post drug treatment 123I SPECT imaging, a treatment according to guidelines for iodine positive lesions will be performed. The follow up of the patients will be conducted as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed radioiodine refractory metastatic thyroid carcinoma of follicular origin (including papillary and its respective variants).
* Confirmation of the mutation status of BRAF gene (primary tumor, recurrent tumor, or metastasis) .
* Patients who do not undergo a systemic treatment with sorafenib or lenvatinib or chemotherapy or with other TKIs or other investigational drugs.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 15 mm with CT scan, MRI, or calipers by clinical exam. Tumors in previously irradiated fields may be considered measureable if there is evidence of tumor progression after radiation treatment.
* RAI-refractory disease on structural imaging, defined as following:

A metastatic lesion that is not radioiodine-avid on a diagnostic or therapeutic radioiodine scan performed less than 1 year prior to enrollment in the current study, There are no size limitations for the index lesion used to satisfy this entry criterion.

* No recent treatment for thyroid cancer as defined as:

  1. No prior 131I therapy is allowed < 6 months prior to initiation of therapy on this protocol. A diagnostic study using < 400 MBq (±100) of 131I is not considered 131I therapy.
  2. No external beam radiation therapy < 4 weeks prior to initiation of therapy on this protocol. (Previous treatment with radiation for any indication is allowed if the investigator judges that the previous radiation does not significantly compromise patient safety on this protocol.)
  3. No chemotherapy or targeted therapy (e.g., tyrosine kinase inhibitor) is allowed < 4 weeks prior to the initiation of therapy on this protocol.
* Age ≥ 18 years
* ECOG performance status ≤ 2.
* Life expectancy of greater than 3 months. Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Patients must have normal organ and bone marrow function as defined below:
* Absolute neutrophil count (ANC) > 1.5x10^9/L
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100 x 10^9/L
* Albumin ≥ 2.5 g/dL
* Total bilirubin ≤ 1.5x institutional ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x institutional ULN unless it is related to the primary disease
* creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) ≥ 50 mL/min OR 24-hour urine creatinine clearance ≥ 50 mL/min
* Negative pregnancy test within 7 days prior to starting the study premenopausal women. Women of non-childbearing potential may be included without pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. Effective methods of contraception are defined as those, which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must agree to undergo to research biopsy of a malignant lesion if the mutation status cannot be proven through archival tissue specimen.
* Availability of archival tumor tissue from the thyroid cancer primary or metastasis (a tissue block or a minimum of 30 unstained slides would be required. Patients with less archival tissue available may still be eligible for the study after discussion with the Principal Investigator). This does not apply to patients who undergo a biopsy.

Exclusion Criteria:

* Concomitant malignancies or previous malignancies of life-limiting potential within the last 3 years.
* Use of other investigational drugs within 28 days preceding the first dose of drug treatment during this study.
* Known leptomeningeal or brain metastases or spinal metastases.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib and/or to dabrafenib or other known contents of the two investigational drugs.
* History or evidence of cardiovascular risk including any of the following:
* History or evidence of current, clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to the initiation of therapy on this protocol are eligible).
* History of acute coronary syndromes (specifically, myocardial infarction and unstable angina), severe/unstable angina, coronary angioplasty, or stenting within 6 months prior to the initiation of therapy on this protocol.
* History of symptomatic congestive heart failure within 6 months prior to the initiation of therapy on this protocol.
* History of cerebrovascular attack or transient ischemic attack within 6 months prior to the initiation of therapy on this protocol.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant, lactating, or breast feeding women.
* Patients unable to follow a low iodine diet or requiring medication with high content in iodide (amiodarone).
* Patients who received iodinated intravenous contrast as part of a radiographic procedure within 3 months of study registration. Those that have had iodinated intravenous contrast within this time frame may still be eligible if a urinary iodine analysis reveals that the excess iodine has been adequately cleared after the last intravenous contrast administration.
* Unwillingness or inability to comply with study and follow-up procedures.
* Disorders of eye background as listed in the respective study drug prescribing information.
* Patients with pancreatitis, prolonged QTc-time on EKG, uncontrolled hypertension, thrombosis or high risk of bleedings.
* Condition of patient which is critical to participate in this study in the discretion of the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with sufficiently increased tumoral iodine incorporation | At the time point of 123I whole-body scintigraphy, 3 weeks after the start of redifferentiation therapy
  To determine the proportion of patients with BRAF WT RAIR thyroid cancer in which trametinib and the proportion of patients with BRAF MUT RAIR thyroid cancer in which the combination-therapy of dabrafenib and trametinib can increase tumoral iodine incorporation sufficiently.

SECONDARY OUTCOMES:
Changes in thyroglobulin levels | Within 12 months after redifferentiation therapy
  Declines or increases in thyroglobulin levels after redifferentiation therapy
The incidence and severity of adverse effects under trametinib (+dabrafenib) treatment | Within 3 months
  The incidence and severity of adverse effects and necessary therapeutic measures are monitored pursuant to CTCAE 4.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang P Fendler, MD, Principal Investigator — Department of Nuclear Medicine, Essen University Hospital
Locations (1):
- Manuel M. Weber, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No